CLINICAL TRIAL: NCT04489914
Title: Observational Study on the Application of High-Flow Therapy in the Postinterventional Follow-up Care of Patients With Percutaneous Interventional Aortic Valve Replacement
Brief Title: Observational Study on the Application of High-Flow Therapy After Percutaneous Transfemoral Aortic Valve Replacement
Status: Completed | Type: Observational
Sponsor: Drägerwerk AG & Co. KGaA (Industry)
Responsible Party: Sponsor
Other Study IDs: TAVI-STAR
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: High-Flow Oxygen Therapy — high-flow oxygen therapy after percutaneous transfemoral aortic valve replacement

SUMMARY:
Percutaneous catheter-assisted valve replacement in aortic position (TAVI) for patients with high perioperative risk has become a standard method in recent years. In addition to the detection of bleeding and cardiac rhythm complications, follow-up care is mainly focused on the monitoring of respiratory parameters after an operation under intubation anesthesia or deep analgosedation. In addition to normal oxygen therapy, non-invasive ventilation and, in case of weaning failure, renewed tracheal intubation in the first 24 h after TAVI have been considered. High flow oxygen therapy (HFOT) now provides a good opportunity to treat patients with a warmed and humidified air-oxygen mixture and to independently control the oxygen content in the inhaled air and the flow in the pharyngeal area.

The aim of the Study is to investigate the Change in oxygenation after high-flow oxygen therapy as a measure of weaning success in postinterventional patients after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* High-flow oxygen therapy after TAVI

Exclusion Criteria:

* patients without consent
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University hospital
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Change of Horovitz index | 24 hours
  The Gradient of paO2/FiO2 will be determined after TAVI via blood gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Graf, Dr, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Schleswig-Holstein, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No